CLINICAL TRIAL: NCT06177496
Title: Influence of Sarcopenia on Mortality and Disease Progression in Hepatocellular Carcinoma Treated With Ablation, Embolization and Sorafenib
Brief Title: Influence of Sarcopenia in Hepatocellular Carcinoma Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelwahab Mohamed, Lecturer of Tropical Medicine and Gastroenterology, Sohag University
Other Study IDs: Soh-Med-23-09-11PD
Record Dates: First submitted 2023-11-27; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: HCC patients underwent local ablation
  Interventions: Procedure: local ablation
- Group B: HCC patients underwent TACE
  Interventions: Procedure: TACE
- Group C: HCC patients received sorafenib
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Procedure: local ablation — treatment of HCC
  Groups: Group A
Procedure: TACE — treatment of HCC
  Groups: Group B
Drug: Sorafenib — treatment of HCC
  Groups: Group C

SUMMARY:
Liver cancer poses a major threat to the global cancer burden, and the number of deaths is estimated to be more than one million annually by 2030. Locoregional therapies such as transarterial chemoembolization (TACE), transarterial radioembolization (TARE), and radiation are associated with improved survival and quality of life for patients with unresectable HCC [Couri and Pillai, 2019]. However, curative therapies or locoregional therapies are not applicable to approximately 50% of HCC cases who are diagnosed at an advanced stage and have progression with transarterial therapies [Park et al., 2015]. For these patients, sorafenib, lenvatinib, and atezolizumab combined with bevacizumab have been approved as the first-line systemic therapy [Fan et al., 2022].

Sarcopenia is a progressive and generalized skeletal muscle disease characterized by accelerated loss of muscle mass and function [Cruz-Jentoft and Sayer, 2019]. It has been associated with higher mortality among the general population and patients with cancer. This study aims to assess the possible role of sarcopenia in predicting the outcome of HCC patients following a variety of treatments including local ablation, TACE and sorafenib.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of hepatocellular carcinoma.
2. Treatment-naive patients who underwent local ablation, TACE or sorafenib as a primary treatment .

Exclusion Criteria:

1. Use of other another HCC treatment modality e.g., resection.
2. Use of combined treatments e.g., simultaneous use of embolic therapy with ablation.
3. Patients with recurrent HCC.
4. Patients with secondaries from extra-hepatic primary tumors.
5. Incomplete data at the diagnosis, treatment or follow up time-points.
6. Loss of patients follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naive hepatocellular carcinoma patients who underwent local ablation, TACE or sorafenib as a primary treatment.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | for at least 1 year from the treatment
  time from treatment till death or last contact

SECONDARY OUTCOMES:
Recurrence-free survival | for at least 1 year from the treatment
  time from HCC treatment to tumor relapse (identified by imaging) or last contact
Progression-free survival | for at least 1 year from the treatment
  time from HCC treatment to tumor progression (identified by imaging) or last contact

IPD SHARING:
Plan to Share IPD: Undecided